CLINICAL TRIAL: NCT02170532
Title: Aerosolized Beta-Agonist Isomers in Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013822
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Levalbuterol; Sodium Chloride

ARMS (5):
- levalbuterol + saline in a breath actuated nebulizer (Active Comparator): 0.5 ml. levalbuterol + 0.5ml saline in a breath actuated nebulizer
  Interventions: Drug: levalbuterol; Drug: saline; Device: breath actuated nebulizer
- levalbuterol + ipratroprium in a breath actuated nebulizer (Active Comparator): 0.5 ml. levalbuterol + 0.5ml ipratroprium in a breath actuated nebulizer
  Interventions: Drug: levalbuterol; Device: breath actuated nebulizer; Drug: ipratroprium
- levalbuterol MDI 2 puffs (Active Comparator): levalbuterol metered dose inhaler 2 puffs
  Interventions: Other: levalbuterol MDI
- levalbuterol MDI + aerochamber max without pause 2 puffs (Active Comparator): levalbuterol MDI + aerochamber max without pause 2 puffs
  Interventions: Other: levalbuterol MDI; Device: aerochamber max
- levalbuterol MDI + aerochamber max with 2 second pause 2 puffs (Active Comparator): levalbuterol MDI + aerochamber max with 2 second pause 2 puffs
  Interventions: Other: levalbuterol MDI; Device: aerochamber max

INTERVENTIONS:
Drug: levalbuterol — 0.5 ml. levalbuterol
  Arms: levalbuterol + ipratroprium in a breath actuated nebulizer; levalbuterol + saline in a breath actuated nebulizer
Drug: saline — 0.5ml saline
  Arms: levalbuterol + saline in a breath actuated nebulizer
Other: levalbuterol MDI
  Arms: levalbuterol MDI + aerochamber max with 2 second pause 2 puffs; levalbuterol MDI + aerochamber max without pause 2 puffs; levalbuterol MDI 2 puffs
Device: breath actuated nebulizer
  Arms: levalbuterol + ipratroprium in a breath actuated nebulizer; levalbuterol + saline in a breath actuated nebulizer
Device: aerochamber max
  Arms: levalbuterol MDI + aerochamber max with 2 second pause 2 puffs; levalbuterol MDI + aerochamber max without pause 2 puffs
Drug: ipratroprium
  Arms: levalbuterol + ipratroprium in a breath actuated nebulizer

SUMMARY:
Dr. MacIntyre and his colleagues are studying inhaled medications in asthma. There are two new medications that have been approved by the United States Food and Drug Administration (FDA): levalbuterol and formoterol. Both of these drugs are similar to standard asthma bronchodilator drugs but offer theoretical advantages in terms of fewer side effects. There are also newer devices to deliver these medications into the lungs: breath actuated nebulizers (BANs) and non-static chambers (Aerochamber-max) that can be used with metered dose inhalers (MDIs or "puffers"). The purpose of this study is to deliver these new medications using several different devices and measuring lung function, heart rate, and sensations of breathlessness.

DETAILED DESCRIPTION:
Patients will be studied on five separate mornings. The duration of the study and frequency of the visits will be solely dependant on the subject availability. Each subject will receive all 5 treatments in the same order.

ELIGIBILITY:
Inclusion Criteria:

* stable mild to moderate persistent asthma as defined by the National Asthma Education and Prevention Program
* greater than 18 years of age
* requiring bronchodilator therapy either routinely or on a as needed (PRN)basis
* stable with respect to respiratory disease and at least four weeks removed from the most recent acute exacerbation of the disease
* patients may or may not be on inhaled corticosteroids

Exclusion Criteria:

* no unstable cardiovascular symptoms
* no unstable angina
* must be at least four weeks removed from an acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacIntyre, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All subjects will receive all 5 treatments on 5 different treatment days. Each subject will receive all 5 treatments in the same order.
Period: Overall Study
Arm/Group | All Subjects
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects will receive all 5 treatments on 5 different treatment days. Each subject will receive all 5 treatments in the same order.
Arm/Group | All Subjects
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants]
  18 & older | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Forced Expiratory Volume at One Second (FEV1)
Time Frame: Baseline (before treatment), 30 minutes, 1, 2, 4, 6, and 8 hours post treatment
Population: The same 10 subjects received each of the 5 treatments in the same order. Subjects 1-5 were not included in 6 and 8 hour time points.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Levalbuterol + Saline in a Breath Actuated Nebulizer: 0.5 ml. levalbuterol + 0.5ml saline in a breath actuated nebulizer
  levalbuterol: 0.5 ml. levalbuterol
  saline: 0.5ml saline
  breath actuated nebulizer
- Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer: 0.5 ml. levalbuterol + 0.5ml ipratroprium in a breath actuated nebulizer
  levalbuterol: 0.5 ml. levalbuterol
  breath actuated nebulizer
  ipratroprium
- Levalbuterol Metered Dose Inhaler (MDI) 2 Puffs: levalbuterol metered dose inhaler (MDI) 2 puffs
  levalbuterol MDI
- Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs: levalbuterol metered-dose inhaler (MDI) + aerochamber max without pause 2 puffs
  levalbuterol MDI
  aerochamber max
- Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs: levalbuterol metered dose inhaler (MDI) + aerochamber max with 2 second pause 2 puffs
  levalbuterol MDI
  aerochamber max
Arm/Group | Levalbuterol + Saline in a Breath Actuated Nebulizer | Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer | Levalbuterol Metered Dose Inhaler (MDI) 2 Puffs | Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs | Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
percentage of change
  30 minutes | 20 (23.19) | 20 (16.55) | 20 (19.85) | 19 (20.64) | 21 (21.10)
  1 hour | 28 (31.45) | 23 (19.24) | 19 (22.57) | 20 (24.23) | 24 (22.62)
  2 hour | 26 (32.23) | 22 (20.64) | 20 (23.02) | 19 (26.25) | 19 (21.47)
  4 hour | 15 (29.05) | 14 (18.89) | 7 (18.99) | 6 (16.88) | 7 (18.51)
  6 hour | 0 (18.9) | 1 (5.23) | -5 (5.98) | 1 (16.05) | -6 (11.68)
  8 hour | 1 (21.26) | 9 (13.10) | -3 (7.91) | 0 (15.54) | -6 (11.55)

2. Secondary Outcome: Change in 8 Hour Area-under-the-curve FEV1
Time Frame: 0 to 8 hours post dose
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Levalbuterol MDI 2 Puffs: levalbuterol metered dose inhaler 2 puffs
  levalbuterol MDI
- Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs: levalbuterol MDI + aerochamber max without pause 2 puffs
  levalbuterol MDI
  aerochamber max
- Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs: levalbuterol MDI + aerochamber max with 2 second pause 2 puffs
  levalbuterol MDI
  aerochamber max
Arm/Group | Levalbuterol + Saline in a Breath Actuated Nebulizer | Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer | Levalbuterol MDI 2 Puffs | Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs | Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
percentage of change | 5450 (7039) | 4729 (4275) | 3893 (4949) | 3805 (5253) | 4195 (4795)

3. Secondary Outcome: Change in Heart Rate
Time Frame: Baseline (before treatment), 30 minutes, 1, 2, 4, 6, and 8 hours post treatment
Population: Data for this outcome measure is not reported because the data was not collected.
Arm/Group | Levalbuterol + Saline in a Breath Actuated Nebulizer | Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer | Levalbuterol MDI 2 Puffs | Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs | Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Tremor Assessment Measured by a Scale
Description: Tremor assessment will be made on outstretched hands (0 = none, 1+ = fine tremor, barely perceptible, 2+ = obvious tremor).
Time Frame: Baseline (before treatment), 30 minutes, 1, 2, 4, 6, and 8 hours post treatment
Population: Data for this outcome measure is not reported because the data was not collected.
Arm/Group | Levalbuterol + Saline in a Breath Actuated Nebulizer | Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer | Levalbuterol MDI 2 Puffs | Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs | Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in Dyspnea Response as Measured by the University of California, San Diego (UCSD) Dyspnea Scale
Time Frame: Baseline (before treatment), 30 minutes, 1, 2, 4, 6, and 8 hours post treatment
Population: Data for this outcome measure is not reported because the data was not collected.
Arm/Group | Levalbuterol + Saline in a Breath Actuated Nebulizer | Levalbuterol + Ipratroprium in a Breath Actuated Nebulizer | Levalbuterol MDI 2 Puffs | Levalbuterol MDI + Aerochamber Max Without Pause 2 Puffs | Levalbuterol MDI + Aerochamber Max With 2 Second Pause 2 Puffs
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes